CLINICAL TRIAL: NCT05919264
Title: A Phase 1/2 Study of FOG-001 in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: FOG-001 in Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Parabilis Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FOG-001-101
Record Dates: First submitted 2023-05-19; First posted 2023-06-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Colorectal Cancer; Solid Tumor; Locally Advanced Solid Tumor; Metastatic Cancer; WNT Pathway; β-catenin; Beta-catenin; Adenomatous Polyposis Coli; APC; HCC; Desmoid; Microsatellite Stable Colorectal Cancer; Metastatic Castration-resistant Prostate Cancer; FAP; Endometrial Carcinoma; Prostate Cancer; Microsatellite Instability-High Colorectal Cancer; CTNNB1; Adamantinomatous Craniopharyngioma
Keywords: Cancer; Solid Tumor; Locally Advanced Solid Tumor; Metastatic Cancer; WNT Pathway Activating Mutation (WPAM); Colorectal Cancer (CRC); Microsatellite Stable (MSS); Desmoid
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Adenomatous Polyposis Coli; Desmoid Tumors; Endometrial Neoplasms; Prostatic Neoplasms; Craniopharyngioma | interventions — Leucovorin; Fluorouracil; Oxaliplatin; Nivolumab; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part 1a (Experimental): Solid Tumors with any WNT-Pathway Activating Mutation (WPAM) or Microsatellite Stable (MSS) Colorectal Cancer (CRC), irrespective of WPAM status
  Interventions: Drug: FOG-001
- Part 1b (Experimental): MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001
- Part 1c (Experimental): Hepatocellular Carcinoma (documented WPAM in APC or CTNNB1 required)
  Interventions: Drug: FOG-001
- Part 1d-1 (Experimental): Desmoid Tumors
  Interventions: Drug: FOG-001
- Part 1d-2 (Experimental): Desmoid Tumors
  Interventions: Drug: FOG-001
- Part 1e-1 (Experimental): Solid Tumors with documented WPAM or MSS CRC, irrespective of WPAM status
  Interventions: Drug: FOG-001
- Part 1e-2 (Experimental): Solid Tumors with documented WPAM or MSS CRC, irrespective of WPAM status
  Interventions: Drug: FOG-001
- Part 1f-1 (Experimental): MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001; Drug: mFOLFOX-6; Drug: Bevacizumab
- Part 1f-2 (Experimental): Solid Tumors with documented WPAM or MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001; Drug: Nivolumab
- Part 1f-3 (Experimental): MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001; Drug: Trifluridine/tipiracil; Drug: Bevacizumab
- Part 2a (Experimental): MSS CRC, irrespective of WPAM status
  Interventions: Drug: FOG-001
- Part 2b (Experimental): Solid Tumors with documented WPAM
  Interventions: Drug: FOG-001
- Part 2c (Experimental): Hepatocellular Carcinoma (documented WPAM in APC or CTNNB1 required)
  Interventions: Drug: FOG-001
- Part 2d (Experimental): Desmoid Tumors
  Interventions: Drug: FOG-001
- Part 2e (Experimental): Metastatic Castration-Resistant Prostate Cancer (documented WPAM in APC or CTNNB1 required)
  Interventions: Drug: FOG-001
- Part 2f-1 (Experimental): MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001; Drug: mFOLFOX-6; Drug: Bevacizumab
- Part 2f-2 (Experimental): Solid Tumors with documented WPAM or MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001; Drug: Nivolumab
- Part 2f-3 (Experimental): MSS CRC (known WPAM negative participants are not eligible)
  Interventions: Drug: FOG-001; Drug: Trifluridine/tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: FOG-001 — FOG-001 will be administered IV at assigned doses in continuous cycles of 28 days
Drug: mFOLFOX-6 — mFOLFOX-6 will be administered per the prescribing information in combination with FOG-001
  Other Names: Leucovorin, 5-fluorouracil, Oxaliplatin
  Arms: Part 1f-1; Part 2f-1
Drug: Nivolumab — Nivolumab will be administered per the prescribing information in combination with FOG-001
  Other Names: Opdivo
  Arms: Part 1f-2; Part 2f-2
Drug: Trifluridine/tipiracil — Trifluridine/tipiracil will be administered per the prescribing information in combination with FOG-001
  Other Names: Lonsurf
  Arms: Part 1f-3; Part 2f-3
Drug: Bevacizumab — Bevacizumab will be administered per the prescribing information in combination with FOG-001
  Other Names: Avastin
  Arms: Part 1f-1; Part 1f-3; Part 2f-1; Part 2f-3

SUMMARY:
The goal of this clinical trial is to determine if FOG-001 is safe and effective in participants with locally advanced or metastatic cancer.

DETAILED DESCRIPTION:
This is a FIH, Phase 1/2, multicenter, open-label, non-randomized, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, pharmacodynamics, and antitumor activity of FOG-001 as monotherapy and in combination with other anticancer agents in participants with advanced or metastatic solid tumors likely or known to have a Wnt pathway activating mutation (WPAM).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ and marrow function.

Additional Inclusion Criteria for Dose Escalation Cohorts (Part 1a and Part 1e):

* Diagnosis of treatment-refractory advanced/metastatic solid tumor that is non-MSI-H or non-dMMR colorectal cancer (CRC) or any other solid tumor with documented WNT- pathway activating mutations (WPAMs).

Additional Inclusion Criteria for Dose Escalation Cohorts (Part 1b):

* Diagnosis of treatment-refractory advanced/metastatic non-MSI-H or non-dMMR CRC.
* At least one lesion that is suitable for a core needle biopsy.

Additional Inclusion Criteria for Dose Escalation and Dose Expansion Cohorts (Part 1c and Part 2c):

* Diagnosis of HCC with a documented WPAM (by local testing) in APC or CTNNB1. HCC that is radiographically confirmed without tissue biopsy may be enrolled with a documented CTNNB1 mutation (e.g., by ctDNA).

Additional Inclusion Criteria for Dose Escalation and Dose Expansion Cohorts (Part 1d and Part 2d):

* Desmoid tumor (aggressive fibromatosis)

Additional Inclusion Criteria for Dose Escalation and Dose Expansion Cohorts (Part 1f-1 and Part 2f-1) FOG-001 + FOLFOX + Bevacizumab:

* Diagnosis of locally advanced or metastatic non-MSI-H or non-dMMR CRC
* Participants with tumors known to be negative for APC LoF mutations or CTNNB1 GoF mutations (per NGS tests) are not eligible.
* One dose of mFOLFOX6 in the unresectable or metastatic setting prior to enrollment is allowed.

Additional Inclusion Criteria for Dose Escalation and Dose Expansion Cohorts (Part 1f-2 and Part 2f-2): FOG-001 + Nivolumab

* Non-MSI-H or non-dMMR (by local testing) CRC with or without liver metastases.
* MSI-H CRC or solid tumors that are WPAM and resistant to a-PD-1/PD-L1
* Participants with tumors known to be negative for APC LoF mutations or CTNNB1 GoF mutations (per NGS tests) are not eligible

Additional Inclusion Criteria for Dose Escalation and Dose Expansion Cohorts (Part 1f-3 and Part 2f-3): FOG-001 + Trifluridine/Tipiracil + Bevacizumab

* Diagnosis of locally advanced or metastatic non-MSI-H or non-dMMR (by local testing) CRC
* Participants with tumors known to be negative for APC LoF mutations or CTNNB1 GoF mutations (per NGS tests) are not eligible.

Additional Inclusion Criteria for Dose Expansion Cohort (Part 2a):

* Diagnosis of locally advanced or metastatic non-MSI-H or non-dMMR (by local testing) CRC

Additional Inclusion Criteria for Dose Expansion Cohort (Part 2b):

* Diagnosis of advanced or metastatic solid tumors with a documented WPAM (by local testing) or equivalent evidence

Exclusion Criteria:

* Known history of bone metastasis. Bone metastasis are allowed for patients with mCRPC.
* Evidence of vertebral compression fracture or non-traumatic bone fracture within the past 12 months and who are not receiving antiresorptive therapy.
* Osteoporosis, which is defined as a T-score of ≤-2.5 at the lumbar spine (L1 - L4), left (or right) femoral neck or left (or right) total hip as determined by DXA scan.
* Uncontrolled inflammatory bowel disease (i.e., ulcerative colitis or Crohn's disease)
* Unstable/inadequate cardiac function.
* Has known meningeal carcinomatosis, leptomeningeal carcinomatosis, spinal cord compression, or symptomatic or unstable brain metastases.
* Pregnant, lactating, or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
During dose escalation and dose expansion measure incidence and severity of treatment emergent adverse events by CTCAE v5.0 | Through study completion, an average of 10 months
  Number and severity of treatment emergent adverse events as assessed by CTCAE v5.0
During dose escalation characterize dose-limiting toxicities (DLTs) | 1 treatment cycle (28 days)
  Incidence of DLTs
During dose expansion describe the Overall Response Rate using RECIST v1.1 | Every 63 days until study completion, approximately 10 months on average
  The rate of objective responses (Partial & Complete) using RECIST v1.1
During dose expansion describe the Disease Control Rate using RECIST v1.1 (Part 2a only) | 4 months
  The rate of objective responses (Stable, Partial, & Complete) using RECIST v1.1
During dose expansion describe the PSA30 response rate for participants with prostate cancer | Baseline, weekly during the first 2 cycles (56 days), bi-weekly during the Cycle 3 (28 days), and then monthly (up to approximately 7 months)
  The response to treatment as a 30% or greater reduction in PSA levels from baseline

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of FOG-001 and associated metabolites | During first 2 cycles (56 days)
Time to achieve Cmax (Tmax) of FOG-001 and associated metabolites in plasma | During first 2 cycles (56 days)
Area under the plasma concentration-time curve (AUC) of FOG-001 and associated metabolites | During first 2 cycles (56 days)
Plasma trough concentration (Ctrough) of FOG-001 and associated metabolites | During first 2 cycles (56 days)
Clearance (CL) of FOG-001 from the plasma | During first 2 cycles (56 days)
Volume of distribution of FOG-001 | During first 2 cycles (56 days)
During dose escalation select the preliminary recommended Phase 2 dose and dosing schedule of study drug | Through Part 1 study completion
Rate of DLTs across dose levels | During Cycle 1 (28 days)
During dose escalation Part 1b to evaluate the pharmacodynamic activity in tumors | During first 2 cycles (56 days)
  Change in tumor Myc expression (on-study compared to baseline)
During dose escalation and expansion to describe Best Overall Response Rate using RECIST v1.1 | Every 63 days until study completion, approximately 10 months on average
  Best response to treatment using RECIST v1.1
During dose escalation and expansion to describe Duration of Response using RECIST v1.1 | Every 63 days until study completion, approximately 10 months on average
  Time from initial objective response (partial response or complete response) to disease progression
During dose escalation and expansion describe Progression Free Survival | From date of randomization until the date of first disease progression, an average of 10 months
  Progression Free Survival (PFS) using RECIST v1.1
During dose escalation and expansion describe the Disease Control Rate using RECIST v1.1 | Every 63 days until study completion, approximately 10 months on average
  The rate of objective responses (Stable, Partial, & Complete) using RECIST v1.1
During dose escalation and expansion describe the Time To Progression using RECIST v1.1 | From date of randomization until the date of first disease progression, an average of 10 months
  Time To Progression (TTP) using RECIST v1.1
During dose escalation and expansion describe radiographic Progression Free Survival for participants with prostate cancer | From date of randomization until the date of first disease progression, an average of 10 months
  Radiographic Progression Free Survival (rPFS) using PCWG3 assessment criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ramos, DO, Study Chair — Parabilis Medicines, Inc.
Locations (23):
- United States (23):
  - Honor Health, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona, Tucson, Arizona
  - Stanford Cancer Institute, Stanford University, Palo Alto, California
  - University of California San Francisco, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Johns Hopkins University, Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Lake Mary, Florida
  - Johns Hopkins University, The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No